CLINICAL TRIAL: NCT01010035
Title: Plasma Kinetics Study of Free Cholesterol and Cholesteryl Ester in Type 2 Diabetes Mellitus Patients
Brief Title: Cholesterol Metabolism and Lipid Transfer in Diabetes
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Antonio Carlos Lerario/ MD, PhD, university of são Paulo
Other Study IDs: LIPIDSDM
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; dyslipidemia; kinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- type 2 diabetes: patients with diagnosis of Type 2 diabetes mellitus
  Interventions: Other: Plasma kinetic study
- Control: non type 2 diabetes mellitus
  Interventions: Other: Plasma kinetic study

INTERVENTIONS:
Other: Plasma kinetic study — this study is done with the injection of LDL-like nanoemulsion doubly labeled with 14C- cholesteryl oleate and 3H- cholesterol, with a total radioactivity injection dose of 0.03mSV. Blood sample collected in a pre established period of time in 24 hours.
  Other Names: LDL-like nanoemulsion

SUMMARY:
The diabetic dyslipidemia is one of the most important risk factor in the development of coronary artery disease. The low density lipoprotein (LDL)-like nanoemulsions is being used to study the clearance of cholesteryl ester and free cholesterol from intravascular in patients with advanced coronary artery disease and it was shown a higher removal of free cholesterol and higher deposit in vases of this patients. The aim of this study is to analyze the plasma kinetics of both forms of cholesterol(free ad esterified) in type 2 diabetes patients without a previous history of cardiovascular disease.

DETAILED DESCRIPTION:
Hypercholesterolemia is not typical of type 2 diabetes mellitus dyslipidemia, but alterations in LDL may occur related to atherogenesis.Cholesterol exist in two main forms in organism: free cholesterol and the esterified cholesterol. An artificial model to study this two forms of cholesterol is the use of LDL-like nanoemulsion doubly labeled with 14C-cholesteryl esters and 3H- cholesterol. This nanoemulsion is made without protein and when in the intravascular compartment it is able to acquires apolipoproteins from others lipoproteins, such apos A's, C's and E. This model allowed us to use the nanoemulsion particle as a probe to study the lipoproteins receptor binding and the cholesterol esterification process.

ELIGIBILITY:
Inclusion Criteria:

* without a previous cardiovascular disease
* if arterial hypertension, or in use of antihypertensive drugs- it must be well controled with a systolic Blood pressure level <130mmHg and diastolic <85mmHg.
* total cholesterol < 6 mmol/L
* LDL- cholesterol <4 mmol/L

Exclusion Criteria:

* use of drugs- statins, fibrates, glucocorticoids, thiazolidinediones
* nephropathy- the presence of microalbuminuria(ratio of microalbuminuria/creatinin >30 ug/mg) or serum creatinin above 98umol/L in woman and above 115 umol/L in man
* retinopathy
* neuropathy presence of chronic disease: heart failure, chronic obstructive pulmonary disease, inflammatory disease and cancer

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient of the endocrinology clinics of Hospital das clinicas of University of São Paulo Medical school
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
to identify the removal of the free and esterified cholesterol in type 2 diabetes patients | day of test

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C Lerario, MD, pHd, Principal Investigator — University of Sao Paulo
Locations (1):
- Endocrinology service and Lipid laboratory of Heart Institute of University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Santos RD, Hueb W, Oliveira AA, Ramires JA, Maranhao RC. Plasma kinetics of a cholesterol-rich emulsion in subjects with or without coronary artery disease. J Lipid Res. 2003 Mar;44(3):464-9. doi: 10.1194/jlr.M200331-JLR200. Epub 2002 Dec 1. PMID 12562871
- [Background] Santos RD, Chacra AP, Morikawa A, Vinagre CC, Maranhao RC. Plasma kinetics of free and esterified cholesterol in familial hypercholesterolemia: effects of simvastatin. Lipids. 2005 Jul;40(7):737-43. doi: 10.1007/s11745-005-1437-6. PMID 16196425
- [Background] Couto RD, Dallan LA, Lisboa LA, Mesquita CH, Vinagre CG, Maranhao RC. Deposition of free cholesterol in the blood vessels of patients with coronary artery disease: a possible novel mechanism for atherogenesis. Lipids. 2007 May;42(5):411-8. doi: 10.1007/s11745-007-3041-9. Epub 2007 Apr 19. PMID 17443358